CLINICAL TRIAL: NCT04091334
Title: Monitoring Patients With Acute Dyspnea With Serial Focused Ultrasound of the Heart and the Lungs
Brief Title: Monitoring Patients With Shortness of Breath With Repeated Ultrasound Examinations
Acronym: MODUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slagelse Hospital (Other)
Collaborators: Odense University Hospital (Other); Holbaek Sygehus (Other); Zealand University Hospital (Other); Horsens Hospital (Other); Herning Hospital (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REG-056-2019
Record Dates: First submitted 2019-09-05; First posted 2019-09-16 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Dyspnea
Keywords: Dyspnea; Ultrasound; Point-of-care; Focused; Serial; Monitoring
MeSH Terms: conditions — Dyspnea | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serial ultrasound group (Experimental): Will received standard care and monitoring and in addition, have focused ultrasound examination of the heart and the lungs done twice.
  The investigator is supposed to titrate the treatment according to the findings on the ultrasound examinations.
  Interventions: Device: Focused ultrasound of the lungs (FLUS) and focused cardiac ultrasound (FoCUS); Other: Standard care
- Standard care group (Active Comparator): Standard care and monitoring.
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Focused ultrasound of the lungs (FLUS) and focused cardiac ultrasound (FoCUS) — FLUS: Scanning 8 zones of the front and lateral of the thorax. Record number of B-lines, consolidations, pneumothorax, pleural effusions.
  FoCUS: Scan the heart in different views and record the ejection fraction, size of the right side of the heart, pericardial effusion, tricuspid annular plane systolic excursion (TAPSE), inferior vena cava (IVC) diameter, and IVC collapsibility Index (IVC-CI).
  Arms: Serial ultrasound group
Other: Standard care — Standard care and evaluation and monitoring

SUMMARY:
Purpose of the study: The purpose of the trial is to investigate whether repeated ultrasound scans of the heart and lungs of patients with shortness of breath may help to optimize their treatment. This patient group is characterized by an extended hospitalization and a high mortality rate. Therefore, it is essential to be able to target the treatment in order to shorten length of stay, prevent readmissions, and improve survival in these patients. Ultrasound scanning used in this way is novel.

The study method: Initially, all patients will receive standard evaluation and ultrasound of the heart and the lungs. Then the patients are randomly assigned into two groups. In one group, patients receive standard assessment and treatment. In the second group, the patients, in addition to standard examination and treatment, receive ultrasound scans of their heart and lungs after two hours and again fire hours after the first scan.

After discharge, the subjects are followed for one year to evaluate what examinations and treatment they received during hospitalization, whether they have been readmitted or died.

DETAILED DESCRIPTION:
Design: Multicenter, randomized, controlled, open-label, and pragmatic trial.

Settings: Several different emergency departments (EDs) in Denmark.

Study flow: After arrival, the patients are screened according to eligibility criteria. If patients meet the inclusion criteria and informed consent is obtained, the patients are randomly assigned to one of two groups. In both groups, the patients received standard evaluation, e.g., blood samples, physical examination, arterial blood gas, and in addition ultrasound examination of the heart and the lungs. In the intervention group, the patients are further examined with serial ultrasound scans of the heart and the lungs after two and four hours after the initial evaluation.

In the course of admittance, the patients will have there baseline characteristics recorded together with the ultrasound findings, symptoms, and vitals. Symptoms will be recorded at a verbal dyspnea symptom scale (VDS) from 0-10.

All data will be registered at the same time points to make comparisons: At 1, 2, 4 and after 5 hours.

Sample size: This is calculated from the primary outcome and with an assumption of a power of 80%, type 1-error of 5%, and 10% dropouts. The calculations are based on previous studies using the VDS on patients with acute dyspnea. The sample size is 103 patients in each group.

Statistical analysis: Baseline characteristics will be summarized and divided into the intervention and control group. Continuous variables will be summarized as means and standard deviation (SD) or medians and interquartile range (IQR) depending on the distribution of the variable. For categorical variables, frequencies and percentages will be reported.

The primary outcome - change in dyspnea on VDS - will be compared between the two groups to detect any difference. Pairwise comparisons of VDS will be made at the same time points in both groups.

The secondary outcomes: Length of stay, death, and the number of readmissions will be compared between the two groups to detect a difference. Time-to-event (dead or readmission) will be visualized with Kaplan Meier curves.

In the case of lost to follow-up or other reasons for missing data both intention-to-treat and per-protocol analysis will be used.

The secondary outcomes in the interventions group: The dynamic changes in inferior vena cava collapsibility index (IVC-CI) and the sum of B-lines will be expressed as means and SD or median and IQR depending on the distribution of the data and compared between the different time points. Furthermore, IVC-CI and the sum of B-lines will be compared to vitals and VDS-score to detect a correlation.

The inter- and intraobserver variability regarding the focused ultrasound will be accessed.

Data management: The registered data on each patient will be recorded and securely stored in an encrypted, logged, and password-protected database called REDCap. All adjustments in the database are logged. The patients are anonymized.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be 18 years or older
* Presented at the ED with shortness of breath (asking the patient upon arrival in the triage what their primary complaint is for a referral to an emergency department)
* Written informed consent obtained from the patient

Exclusion Criteria:

* Patients with dyspnea primary admitted because of a trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
Change in dyspnea severity on a verbal dyspnea scale (VDS) from 0-10 | Assessed within 1 hour from arrival, again after two, four hours and five hours
  Self reported severity of dyspnea. 0 = no dyspnea. 10 = worst dyspnea ever.

SECONDARY OUTCOMES:
Lenght of stay | Assessed after 30 days from inclusion of the last patient.
  Number of days the patients is admitted.
Number of readmission(s) | Assessed up to 12 months from inclusion of the last patient.
  Number of times the patients is readmitted after discharge.
In-hospital all-cause mortality | Assessed after 30 days from inclusion of the last patient.
  Number of patients who dies under the admission
All-cause mortality after discharge | Assessed up to 12 months from inclusion of the last patient.
  Number of patients who dies after discharge.
IVC-CI (inferior vena cava collapsibility index) correlated to vital signs and VDS | Assessed within 1 hour from arrival, again after two, four hours and five hours
B-line count correlated to vital signs and VDS | Assessed within 1 hour from arrival, again after two, four hours and five hours
The changes in IVC-CI between the ultrasound examinations | Assessed within 1 hour from arrival, again after two, four hours and five hours
The changes in B-line count between the ultrasound examinations | Assessed within 1 hour from arrival, again after two, four hours and five hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael D. Arvig, MD, Principal Investigator — Dept. of Emergency Medicine, Slagelse Hospital
Locations (2):
- Denmark (2):
  - Department of Emergency Medicine, Slagelse, Region Sjælland
  - Department of Emergency Medicine, Horsens

IPD SHARING:
Plan to Share IPD: Yes
Raw data (deidentified participant data) may be made available upon request to the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available within 6 months from the completion of the trial.
Access Criteria: Data can be made available if data sharing is in accordance with applicable legislation on the processing of personal data (The General Data Protection Regulation (GDPR)) and Danish Act on Data Protection. Data will be provided through a secured mailing address. Data can only be reused after acceptance from the project manager.

REFERENCES:
- [Background] Mockel M, Searle J, Muller R, Slagman A, Storchmann H, Oestereich P, Wyrwich W, Ale-Abaei A, Vollert JO, Koch M, Somasundaram R. Chief complaints in medical emergencies: do they relate to underlying disease and outcome? The Charite Emergency Medicine Study (CHARITEM). Eur J Emerg Med. 2013 Apr;20(2):103-8. doi: 10.1097/MEJ.0b013e328351e609. PMID 22387754
- [Background] Ray P, Birolleau S, Lefort Y, Becquemin MH, Beigelman C, Isnard R, Teixeira A, Arthaud M, Riou B, Boddaert J. Acute respiratory failure in the elderly: etiology, emergency diagnosis and prognosis. Crit Care. 2006;10(3):R82. doi: 10.1186/cc4926. Epub 2006 May 24. PMID 16723034
- [Background] Lindskou TA, Pilgaard L, Sovso MB, Klojgard TA, Larsen TM, Jensen FB, Weinrich UM, Christensen EF. Symptom, diagnosis and mortality among respiratory emergency medical service patients. PLoS One. 2019 Feb 28;14(2):e0213145. doi: 10.1371/journal.pone.0213145. eCollection 2019. PMID 30817792
- [Background] Gheorghiade M, Follath F, Ponikowski P, Barsuk JH, Blair JE, Cleland JG, Dickstein K, Drazner MH, Fonarow GC, Jaarsma T, Jondeau G, Sendon JL, Mebazaa A, Metra M, Nieminen M, Pang PS, Seferovic P, Stevenson LW, van Veldhuisen DJ, Zannad F, Anker SD, Rhodes A, McMurray JJ, Filippatos G; European Society of Cardiology; European Society of Intensive Care Medicine. Assessing and grading congestion in acute heart failure: a scientific statement from the acute heart failure committee of the heart failure association of the European Society of Cardiology and endorsed by the European Society of Intensive Care Medicine. Eur J Heart Fail. 2010 May;12(5):423-33. doi: 10.1093/eurjhf/hfq045. Epub 2010 Mar 30. PMID 20354029
- [Background] Pivetta E, Goffi A, Lupia E, Tizzani M, Porrino G, Ferreri E, Volpicelli G, Balzaretti P, Banderali A, Iacobucci A, Locatelli S, Casoli G, Stone MB, Maule MM, Baldi I, Merletti F, Cibinel GA, Baron P, Battista S, Buonafede G, Busso V, Conterno A, Del Rizzo P, Ferrera P, Pecetto PF, Moiraghi C, Morello F, Steri F, Ciccone G, Calasso C, Caserta MA, Civita M, Condo' C, D'Alessandro V, Del Colle S, Ferrero S, Griot G, Laurita E, Lazzero A, Lo Curto F, Michelazzo M, Nicosia V, Palmari N, Ricchiardi A, Rolfo A, Rostagno R, Bar F, Boero E, Frascisco M, Micossi I, Mussa A, Stefanone V, Agricola R, Cordero G, Corradi F, Runzo C, Soragna A, Sciullo D, Vercillo D, Allione A, Artana N, Corsini F, Dutto L, Lauria G, Morgillo T, Tartaglino B, Bergandi D, Cassetta I, Masera C, Garrone M, Ghiselli G, Ausiello L, Barutta L, Bernardi E, Bono A, Forno D, Lamorte A, Lison D, Lorenzati B, Maggio E, Masi I, Maggiorotto M, Novelli G, Panero F, Perotto M, Ravazzoli M, Saglio E, Soardo F, Tizzani A, Tizzani P, Tullio M, Ulla M, Romagnoli E; SIMEU Group for Lung Ultrasound in the Emergency Department in Piedmont. Lung Ultrasound-Implemented Diagnosis of Acute Decompensated Heart Failure in the ED: A SIMEU Multicenter Study. Chest. 2015 Jul;148(1):202-210. doi: 10.1378/chest.14-2608. PMID 25654562
- [Background] Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation; American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Oct 15;62(16):e147-239. doi: 10.1016/j.jacc.2013.05.019. Epub 2013 Jun 5. No abstract available. PMID 23747642
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P. 2016 ESC Guidelines for the Diagnosis and Treatment of Acute and Chronic Heart Failure. Rev Esp Cardiol (Engl Ed). 2016 Dec;69(12):1167. doi: 10.1016/j.rec.2016.11.005. No abstract available. English, Spanish. PMID 27894487
- [Background] Gargani L, Volpicelli G. How I do it: lung ultrasound. Cardiovasc Ultrasound. 2014 Jul 4;12:25. doi: 10.1186/1476-7120-12-25. PMID 24993976
- [Background] Volpicelli G, Elbarbary M, Blaivas M, Lichtenstein DA, Mathis G, Kirkpatrick AW, Melniker L, Gargani L, Noble VE, Via G, Dean A, Tsung JW, Soldati G, Copetti R, Bouhemad B, Reissig A, Agricola E, Rouby JJ, Arbelot C, Liteplo A, Sargsyan A, Silva F, Hoppmann R, Breitkreutz R, Seibel A, Neri L, Storti E, Petrovic T; International Liaison Committee on Lung Ultrasound (ILC-LUS) for International Consensus Conference on Lung Ultrasound (ICC-LUS). International evidence-based recommendations for point-of-care lung ultrasound. Intensive Care Med. 2012 Apr;38(4):577-91. doi: 10.1007/s00134-012-2513-4. Epub 2012 Mar 6. PMID 22392031
- [Background] Kelly N, Esteve R, Papadimos TJ, Sharpe RP, Keeney SA, DeQuevedo R, Portner M, Bahner DP, Stawicki SP. Clinician-performed ultrasound in hemodynamic and cardiac assessment: a synopsis of current indications and limitations. Eur J Trauma Emerg Surg. 2015 Oct;41(5):469-80. doi: 10.1007/s00068-014-0492-6. Epub 2015 Jan 8. PMID 26038013
- [Background] Gaskamp M, Blubaugh M, McCarthy LH, Scheid DC. Can Bedside Ultrasound Inferior Vena Cava Measurements Accurately Diagnose Congestive Heart Failure in the Emergency Department? A Clin-IQ. J Patient Cent Res Rev. 2016 Fall-Winter;3(4):230-234. Epub 2016 Nov 11. PMID 27857946
- [Background] Blehar DJ, Dickman E, Gaspari R. Identification of congestive heart failure via respiratory variation of inferior vena cava diameter. Am J Emerg Med. 2009 Jan;27(1):71-75. doi: 10.1016/j.ajem.2008.01.002. PMID 19041537
- [Background] Volpicelli G, Caramello V, Cardinale L, Mussa A, Bar F, Frascisco MF. Bedside ultrasound of the lung for the monitoring of acute decompensated heart failure. Am J Emerg Med. 2008 Jun;26(5):585-91. doi: 10.1016/j.ajem.2007.09.014. PMID 18534289
- [Background] Via G, Storti E, Gulati G, Neri L, Mojoli F, Braschi A. Lung ultrasound in the ICU: from diagnostic instrument to respiratory monitoring tool. Minerva Anestesiol. 2012 Nov;78(11):1282-96. Epub 2012 Aug 3. PMID 22858877
- [Background] Martindale JL. Resolution of sonographic B-lines as a measure of pulmonary decongestion in acute heart failure. Am J Emerg Med. 2016 Jun;34(6):1129-32. doi: 10.1016/j.ajem.2016.03.043. Epub 2016 Mar 19. PMID 27061502
- [Background] Ramasubbu K, Deswal A, Chan W, Aguilar D, Bozkurt B. Echocardiographic changes during treatment of acute decompensated heart failure: insights from the ESCAPE trial. J Card Fail. 2012 Oct;18(10):792-8. doi: 10.1016/j.cardfail.2012.08.358. PMID 23040115
- [Background] Asahi T, Nakata M, Higa N, Manita M, Tabata K, Shimabukuro M. Respiratory Collapse of the Inferior Vena Cava Reflects Volume Shift and Subsequent Fluid Refill in Acute Heart Failure Syndrome. Circ J. 2016 Apr 25;80(5):1171-7. doi: 10.1253/circj.CJ-15-1374. Epub 2016 Mar 29. PMID 27026172
- [Background] Ferrada P, Evans D, Wolfe L, Anand RJ, Vanguri P, Mayglothling J, Whelan J, Malhotra A, Goldberg S, Duane T, Aboutanos M, Ivatury RR. Findings of a randomized controlled trial using limited transthoracic echocardiogram (LTTE) as a hemodynamic monitoring tool in the trauma bay. J Trauma Acute Care Surg. 2014 Jan;76(1):31-7; discussion 37-8. doi: 10.1097/TA.0b013e3182a74ad9. PMID 24368354
- [Background] Yavasi O, Unluer EE, Kayayurt K, Ekinci S, Saglam C, Surum N, Koseoglu MH, Yesil M. Monitoring the response to treatment of acute heart failure patients by ultrasonographic inferior vena cava collapsibility index. Am J Emerg Med. 2014 May;32(5):403-7. doi: 10.1016/j.ajem.2013.12.046. Epub 2014 Jan 3. PMID 24629744
- [Background] Tchernodrinski S, Lucas BP, Athavale A, Candotti C, Margeta B, Katz A, Kumapley R. Inferior vena cava diameter change after intravenous furosemide in patients diagnosed with acute decompensated heart failure. J Clin Ultrasound. 2015 Mar;43(3):187-93. doi: 10.1002/jcu.22173. Epub 2014 Jun 4. PMID 24897939
- [Background] Gargani L, Pang PS, Frassi F, Miglioranza MH, Dini FL, Landi P, Picano E. Persistent pulmonary congestion before discharge predicts rehospitalization in heart failure: a lung ultrasound study. Cardiovasc Ultrasound. 2015 Sep 4;13:40. doi: 10.1186/s12947-015-0033-4. PMID 26337295
- [Background] Spevack R, Al Shukairi M, Jayaraman D, Dankoff J, Rudski L, Lipes J. Serial lung and IVC ultrasound in the assessment of congestive heart failure. Crit Ultrasound J. 2017 Dec;9(1):7. doi: 10.1186/s13089-017-0062-3. Epub 2017 Mar 7. PMID 28271386
- [Background] Saracino A, Weiland TJ, Jolly B, Dent AW. Verbal dyspnoea score predicts emergency department departure status in patients with shortness of breath. Emerg Med Australas. 2010 Feb;22(1):21-9. doi: 10.1111/j.1742-6723.2009.01254.x. Epub 2010 Feb 4. PMID 20136641
- [Background] Saracino A, Weiland T, Dent A, Jolly B. Validation of a verbal dyspnoea rating scale in the emergency department. Emerg Med Australas. 2008 Dec;20(6):475-81. doi: 10.1111/j.1742-6723.2008.01132.x. PMID 19125825
- [Background] Via G, Hussain A, Wells M, Reardon R, ElBarbary M, Noble VE, Tsung JW, Neskovic AN, Price S, Oren-Grinberg A, Liteplo A, Cordioli R, Naqvi N, Rola P, Poelaert J, Gulic TG, Sloth E, Labovitz A, Kimura B, Breitkreutz R, Masani N, Bowra J, Talmor D, Guarracino F, Goudie A, Xiaoting W, Chawla R, Galderisi M, Blaivas M, Petrovic T, Storti E, Neri L, Melniker L; International Liaison Committee on Focused Cardiac UltraSound (ILC-FoCUS); International Conference on Focused Cardiac UltraSound (IC-FoCUS). International evidence-based recommendations for focused cardiac ultrasound. J Am Soc Echocardiogr. 2014 Jul;27(7):683.e1-683.e33. doi: 10.1016/j.echo.2014.05.001. PMID 24951446
- [Derived] Arvig MD, Lassen AT, Gaede PH, Gartner SW, Falster C, Skov IR, Petersen HO, Posth S, Laursen CB. Impact of serial cardiopulmonary point-of-care ultrasound exams in patients with acute dyspnoea: a randomised, controlled trial. Emerg Med J. 2023 Oct;40(10):700-707. doi: 10.1136/emermed-2022-212694. Epub 2023 Aug 18. PMID 37595984
- [Derived] Arvig MD, Lassen AT, Gaede PH, Laursen CB. Monitoring patients with acute dyspnoea with a serial focused ultrasound of the heart and the lungs (MODUS): a protocol for a multicentre, randomised, open-label, pragmatic and controlled trial. BMJ Open. 2020 Jun 3;10(6):e034373. doi: 10.1136/bmjopen-2019-034373. PMID 32499263